CLINICAL TRIAL: NCT04986475
Title: The Effect of Music Therapy on High Risk Pregnant Women of Non-Stress Test and Anxiety Levels
Brief Title: Music Therapy on High Risk Pregnant Women of Non-Stress Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Yasemin ERKAL AKSOY, Lecturer Dr, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12345
Record Dates: First submitted 2021-07-08; First posted 2021-08-02 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Anxiety; Fetal Distress; Music
Keywords: Anxiety; Fetal Distress; High Risk Pregnancy
MeSH Terms: conditions — Anxiety Disorders; Fetal Distress | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In order to ensure randomization in the study, a random numbers table was created by dividing them into two groups based on the number determined on the site https://www.randomizer.org/. In order to prevent bias, in order to divide the women into groups according to the randomization list, the groups were written and sealed in two separate opaque envelopes as intervention (the ney sound is played during the NST procedure) and control (the routine NST procedure was applied). Double blinding was done on request.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Music therapy was applied during the non-stress test.
  Interventions: Other: Music Therapy
- Control (No Intervention): A routine non-stress test was performed.

INTERVENTIONS:
Other: Music Therapy — Music therapy was performed by listening to the ney sound during the non-stress test procedure.
  Arms: Music Therapy

SUMMARY:
Non-stress testing (NST) is one of the most commonly used methods to assess fetal health in the prenatal period because it is an easily interpreted, non-invasive, painless, and short-term diagnostic method. Although NST is a non-invasive and painless diagnostic method, pregnant women may feel anxiety during the procedure.

It is supported by studies that listening to music causes relaxation and reducing anxiety. Therefore, the use of music as a non-pharmacological practice will increase the quality of care of individuals. There are many studies suggesting that music reduces anxiety in low-risk pregnancies during NST application. Different instruments such as ney, rebab, kopuz, dombra are used in Turkish music. In particular, ney has come to the fore in music therapy. The ney, which has different types in history, is an instrument that is closest to the human voice. In a compilation about the music used in music therapy in Turkey, it was stated that there are many social and health studies made with the sound of ney. Determining the effect of music on NST and anxiety in high-risk pregnant women will contribute to the literature.

DETAILED DESCRIPTION:
Non-stress testing (NST) is one of the most commonly used methods to assess fetal health in the prenatal period because it is an easily interpreted, non-invasive, painless, and short-term diagnostic method. Although NST is a non-invasive and painless diagnostic method, pregnant women may feel anxiety during the procedure.

It is supported by studies that listening to music causes relaxation and reducing anxiety. Therefore, the use of music as a non-pharmacological practice will increase the quality of care of individuals. There are many studies suggesting that music reduces anxiety in low-risk pregnancies during NST application. Different instruments such as ney, rebab, kopuz, dombra are used in Turkish music. In particular, ney has come to the fore in music therapy. The ney, which has different types in history, is an instrument that is closest to the human voice. In a compilation about the music used in music therapy in Turkey, it was stated that there are many social and health studies made with the sound of ney. Determining the effect of music on NST and anxiety in high-risk pregnant women will contribute to the literature.

The aim of this study is to determine the effect of music therapy on NST and anxiety levels in high-risk pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Those diagnosed with high-risk pregnancy by a physician (pregnancy-induced hypertension, preeclampsia, eclampsia, gestational diabetes, premature rupture of membranes, pregnancy large or small for gestational age, intrauterine growth retardation, pain/contraction, oligohydramnios, premature birth threat, maternal age 35 age and above, maternal body mass index over 30 (obesity))
* Speaking and understanding Turkish
* Pregnant women with a single fetus
* 32-41 weeks of pregnancy

Exclusion Criteria:

* having twin pregnancy
* with heart disease,
* fetal distress,
* having a fetus with anomaly,
* hereditary anemia,
* pregnant women with sexually transmitted diseases

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants are pregnant women.
Enrollment: 116 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Non stress test evaluation form | up to one hour
  It was created by researchers in order to record and evaluate the findings related to the NST procedure. In the NST evaluation form, fetal heart rate and variability, which were followed for at least 20 minutes, number of accelerations, decelerations and fetal movements, test result (reactive or nonreactive) were included.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI)-Questionnaire | up to one hour
  STAI was used to measure the anxiety level of pregnant women. It was developed by Spielberger et al. (Spielberger et al., 1970) and Öner and Le Compte conducted a Turkish validity and reliability study of the scale (Öner & LeCompte, 1983). In the scale, individuals are provided to express their feelings with 40 expressions. With the state anxiety scale, it is possible to determine how the individual feels at the moment and in the conditions, and with the trait anxiety scale, how he feels outside of the current situation and conditions. The scale is a 4-point Likert type.The last score obtained shows the anxiety level of the individual. High scores from the scale indicate an increased level of anxiety, low scores indicate a decrease.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF

REFERENCES:
- [Background] Şimşek Küçükkelepçe D, Timur Taşhan S. The effect of music on the results of a non-stress test: A non-randomized controlled clinical trial. European Journal of Integrative Medicine [Internet]. 2018 Feb;18:8-12. Available from: https://linkinghub.elsevier.com/retrieve/pii/S1876382018300106
- [Background] Aluş Tokat M. During Pregnancy and Birth of Electronic Fetal Follow. İstanbul: Deomed Press; 2013. 23-62 p.
- [Background] Dönmez S, Dağ H, Kazandı M. The Determination of Pregnant Women's Anxiety and Depression Risk Levels Before Amniocentesis. Acıbadem Üniversitesi Sağlık Bilimleri Dergisi. 2012;3(4):255-61.
- [Background] Muller MA, Bleker OP, Bonsel GJ, Bilardo CM. Nuchal translucency screening and anxiety levels in pregnancy and puerperium. Ultrasound Obstet Gynecol. 2006 Apr;27(4):357-61. doi: 10.1002/uog.2761. PMID 16565991
- [Background] Kafali H, Derbent A, Keskin E, Simavli S, Gozdemir E. Effect of maternal anxiety and music on fetal movements and fetal heart rate patterns. J Matern Fetal Neonatal Med. 2011 Mar;24(3):461-4. doi: 10.3109/14767058.2010.501122. Epub 2010 Jul 7. PMID 20608798